CLINICAL TRIAL: NCT04895709
Title: A Phase 1/2 Study of BMS-986340 as Monotherapy and in Combination With Nivolumab or Docetaxel in Participants With Advanced Solid Tumors
Brief Title: A Study of BMS-986340 as Monotherapy and in Combination With Nivolumab or Docetaxel in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA052-002; 2023-503651-10 (Other: EU CTR); U1111-1265-4508 (Other: WHO)
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Gastric/Gastroesophageal Junction Adenocarcinoma; Microsatellite Stable Colorectal Cancer; Non-Small-Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Urothelial Carcinoma; Pancreatic Adenocarcinoma; Melanoma; Ovarian Neoplasms; Triple Negative Breast Neoplasms
Keywords: BMS-986340; Cervical Cancer; CRC; First-in-human; GEJ; Gastric/Gastroesophageal Junction Adenocarcinoma; HNSCC; Microsatellite Stable Colorectal Cancer; MSS CRC; Nivolumab; Non-Small-Cell Lung Cancer; NSCLC; SCCHN; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Urothelial Carcinoma; Pancreatic Adenocarcinoma; Melanoma; Ovarian Neoplasms; Triple Negative Breast Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Melanoma; Ovarian Neoplasms; Triple Negative Breast Neoplasms | interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1A: BMS-986340 Dose Escalation (Experimental)
  Interventions: Drug: BMS-986340
- Part 2A: BMS-986340 Dose Expansion (Experimental)
  Interventions: Drug: BMS-986340
- Part 1B: BMS-986340 + Nivolumab Dose Escalation (Experimental)
  Interventions: Drug: BMS-986340; Drug: BMS-936558-01
- Part 2B: BMS-986340 + Nivolumab Dose Expansion (Experimental)
  Interventions: Drug: BMS-986340; Drug: BMS-936558-01
- Part 1C: BMS-986340 + Docetaxel Dose Escalation (Experimental)
  Interventions: Drug: BMS-986340; Drug: Docetaxel
- Part 1A-J: BMS-986340 Dose Escalation (Experimental)
  Interventions: Drug: BMS-986340
- Part 1B-J: BMS-986340 + Nivolumab Dose Escalation (Experimental)
  Interventions: Drug: BMS-986340; Drug: BMS-936558-01

INTERVENTIONS:
Drug: BMS-986340 — Specified dose on specified days
Drug: BMS-936558-01 — Specified dose on specified days
  Other Names: Nivolumab
  Arms: Part 1B-J: BMS-986340 + Nivolumab Dose Escalation; Part 1B: BMS-986340 + Nivolumab Dose Escalation; Part 2B: BMS-986340 + Nivolumab Dose Expansion
Drug: Docetaxel — Specified dose on specified days
  Arms: Part 1C: BMS-986340 + Docetaxel Dose Escalation

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and recommended dose(s) of BMS-986340 as monotherapy and in combination with nivolumab or docetaxel in participants with advanced solid tumors. This study is a first-in-human (FIH) study of BMS-986340 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Fresh pre-treatment and on-treatment tumor biopsy must be provided for biomarker analysis.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and at least 1 lesion accessible for biopsy. Fine needle biopsy, cytology, and bone lesion biopsies are not acceptable.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Radiographically documented progressive disease on or after the most recent therapy.
* Received standard-of-care therapies, (except for Part 1C, where participants with prior docetaxel use for the advanced/metastatic setting will be excluded), including an available programmed death (ligand)-1 inhibitor known to be effective in the tumor type for which they are being evaluated.
* Advanced or metastatic disease and have received, be refractory to, not be a candidate for, or be intolerant of existing therapies known to provide clinical benefit for the condition of the participant.

Exclusion Criteria

* Women who are pregnant or breastfeeding.
* Primary central nervous system (CNS) malignancy.
* Untreated CNS metastases.
* Leptomeningeal metastases.
* Concurrent malignancy requiring treatment or history of prior malignancy active within 2 years prior to the first dose of study treatment.
* Active, known, or suspected autoimmune disease.
* Condition requiring systemic treatment with either corticosteroids within 14 days or other immunosuppressive medications within 30 days of the first dose of study treatment.
* Prior organ or tissue allograft.
* Uncontrolled or significant cardiovascular disease.
* Major surgery within 4 weeks of study drug administration.
* History of or with active interstitial lung disease or pulmonary fibrosis.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 949 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2028-07-07 (Estimated); Study Completion 2028-07-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 120 weeks
Incidence of serious adverse events (SAEs) | Up to 120 weeks
Incidence of AEs meeting protocol defined dose-limiting toxicity (DLT) criteria | Up to 120 weeks
Incidence of AEs leading to discontinuation | Up to 120 weeks
Incidence of AEs leading to death | Up to 120 weeks

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of BMS-986340 administered as monotherapy: Maximum concentration (Cmax) | Up to 120 weeks
PK parameters of BMS-986340 administered as monotherapy: Time to maximum concentration (Tmax) | Up to 120 weeks
PK parameters of BMS-986340 administered as monotherapy: Area under the concentration-time curve 1 dosing interval (AUC (TAU)) | Up to 120 weeks
PK parameters of BMS-986340 administered as monotherapy: Observed concentration at the end of the dosing interval (Ctau) | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with nivolumab: Maximum concentration (Cmax) | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with docetaxel: Cmax | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with nivolumab: Time to maximum concentration (Tmax) | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with docetaxel: Tmax | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with nivolumab: Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with docetaxel: AUC(TAU) | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with nivolumab: Observed concentration at the end of the dosing interval (Ctau) | Up to 120 weeks
PK parameters of BMS-986340 administered in combination with docetaxel: Ctau | Up to 120 weeks
Incidence of anti-drug antibodies to BMS- 986340 when administered as monotherapy | Up to 120 weeks
Incidence of anti-drug antibodies to BMS- 986340 when administered in combination with nivolumab | Up to 120 weeks
Incidence of anti-drug antibodies to BMS- 986340 when administered in combination with docetaxel | Up to 120 weeks
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by investigator | At 6 months, 12 months
Disease control rate (DCR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by investigator | At 6 months, 12 months
Duration of response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by investigator | At 6 months, 12 months
Progression-free survival rate (PFSR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by investigator | At 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (50):
- United States (11):
  - Community Cancer Institute, Clovis, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Local Institution - 0062, Iowa City, Iowa
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Local Institution - 0006, New York, New York
  - Local Institution - 0002, New York, New York
  - Local Institution - 0001, Portland, Oregon
  - Local Institution - 0063, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
- Australia (6):
  - Blacktown Hospital, Blacktown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Cabrini Hospital - Malvern, Malvern, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - One Clinical Research, Nedlands, Western Australia
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Hamilton Health Sciences-Juravinski Cancer Centre, Hamilton, Ontario
  - Local Institution - 0009, Toronto, Ontario
  - Centre Hospitalier de luniversite de Montreal, Montreal, Quebec
  - The Ottawa Hospital Cancer Centre, Ottawa
- China (3):
  - Local Institution - 0067, Beijing, Beijing Municipality
  - Local Institution - 0066, Jinan, Shandong
  - Local Institution - 0065, Hangzhou, Zhejiang
- Germany (5):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Carl Gustav Carus Dresden-University Cancer Center Early Clinical Trial Unit, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitaetsklinikum Wuerzburg, Würzburg
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - Local Institution - 0035, Ramat Gan, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Italy (6):
  - Humanitas, Rozzano, Milano
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - ospedale le scotte-U.O.C. Immunoterapia Oncologica, Siena
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan
- Spain (7):
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Institut Catalan d Oncologia (ICO) - Badalona, Badalona, Barcelona [Barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Fundación Jiménez Díaz-START Madrid-FJD, Madrid
  - Centro Integral Oncologico Clara Campal-Hospital HM Universitario Sanchinarro-START Madrid-CIOCC, Madrid
  - Clinica Universidad de Navarra-oNCOLOGY, Pamplona

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04895709.html